CLINICAL TRIAL: NCT03249194
Title: Hepatitis C Virus Donor Positive Kidney Transplantation for Hepatitis C Virus Negative Recipients: A Trial of Ultra-short Duration Direct Acting Anti-viral Prophylaxis To Prevent Virus Transmission From Hepatitis C Viremic Donors To Hepatitis C Negative Kidney Transplant Recipients (DAPPER)
Brief Title: Hepatitis C Virus Donor Positive Kidney Transplantation for Hepatitis C Virus Negative Recipients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20010320
Record Dates: First submitted 2017-08-09; First posted 2017-08-15 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Kidney Transplant; Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — elbasvir-grazoprevir drug combination; sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- HCV+ Donor Kidney Recipient (Experimental): All HCV- participants who receive an HCV+ donor kidney transplant will receive a first 'on-call' dose of Epclusa (sofosbuvir/velpatasvir; Gilead) and then three more doses on post-operative Day 1, 2 and 3. Donor HCV Genotype data will be available by Day 7 of transplant.
  Patients will then be followed by serial HCV PCRs. Patients who are HCV PCR positive by Day 14 will be treated with Epclusa once daily x 12 weeks.
  Interventions: Drug: Direct acting Anti-Viral Therapy using Epclusa or Zepatier

INTERVENTIONS:
Drug: Direct acting Anti-Viral Therapy using Epclusa or Zepatier — All patients will receive one 'on-call' dose of SOFOSBUVIR/VELPATASVIR (Epclusa, Gilead) immediately prior to transplant and one dose on post-operative Day 1 post-transplant. Patients who develop detectable HCV viremia will be initiated on Direct Acting Anti-viral (DAA) therapy between 2-4 weeks post-transplant. Patients with GT1 will be treated with ELBASVIR/GRAZOPREVIR (Zepatier, Merck) and those with GT2 or 3 will be treated with SOFOSBUVIR/VELPATASVIR (Epclusa, Gilead) based upon donor genotyping results
  Other Names: Epclusa, Zepatier

SUMMARY:
The development of direct acting anti-virals (DAAs) for the treatment of Hepatitis C virus (HCV) has changed the landscape of HCV therapy dramatically in the last several years with reported sustained virologic response (SVR) rates in excess of 95% for treatment-naïve HCV positive patients including those who have received liver or kidney transplants. Since these new regimens do not include interferon and have already been studied in the post-liver and kidney transplant setting, they now offer a unique opportunity to expand the donor pool and improve the lives of those awaiting renal transplant. The address this gap in knowledge, the investigators hypothesize that pre-emptive treatment with a direct acting anti-viral HCV medication to cure HCV soon after transplant would allow for safe transplantation of HCV positive kidneys in disadvantaged and needy HCV negative kidney recipients with acceptable risks and improved survivals compared with historical cohorts.

DETAILED DESCRIPTION:
Traditionally, HCV+ kidneys are not offered to HCV- patients on the waiting list. The primary concern with offering HCV+ kidneys to HCV- recipients is a risk of viral transmission. Although data about the long-term impact of HCV+ kidney transplantation in to HCV- recipients is unclear, there was a clear suggestion of an increased risk of liver disease in these patients based upon studies performed in the 1990s. Traditional therapy with Interferon could not be offered to these patients as it can lead of rejection if kidney transplant. It was recently reported that nearly 65% (out of a total 6546) of all HCV+ kidneys were discarded between the years 2005-2014. These kidneys were otherwise of excellent quality and could have benefitted more than 4000 patients with 12,000 plus years of graft life.

Since the recent FDA approval of Direct Acting Anti-virals (DAA), these drugs have now been shown to be safe and efficacious even in the setting of kidney transplant. They could offer a unique opportunity to expand the kidney donor pool. For this study, the investigators hypothesize that pre-emptive treatment with a direct acting anti-viral HCV medication to cure HCV soon after transplant would allow for safe transplantation of HCV+ kidneys in disadvantaged and needy HCV- kidney recipients with acceptable risks and improved survivals compared with historical cohorts. This novel study will develop pilot data on the safety and efficacy of utilizing HCV+ kidneys in high-risk HCV- recipients in order to expand the donor pool and reduce the morbidity and mortality of hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* No evidence of HCV infection by HCV PCR (done at the time of the initial consent)
* Age>60 yrs with an expected waiting time>2 years; or
* Age<60 yrs with any one of the following risk factors: Diabetes, coronary artery disease, peripheral artery disease and/or cerebrovascular disease
* Willingness to provide informed consent
* Absence of a living donor.

Exclusion Criteria:

* Estimated life expectancy of less than one year based on clinical judgment of the investigator
* Prior liver or renal transplantation
* Pregnant women
* Incarcerated patients
* Medical or social condition which in the opinion of the investigator will interfere with or prevent follow-up per protocol
* Unable or unwilling to return for follow-up visits

Donor Exclusion Criteria:

* HBV sAg positive
* HIV PCR or antibody positive
* HCV RNA negative

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Sustained Virologic Response (SVR) | 12 weeks
  Among the patients who develop HCV viremia SVR rates with DAA will be measured
Graft and Patient Survival | 1 year
  Age and co-morbidity will matched historical HCV- recipients as controls. Patient survival will also be compared to a contemporary cohort of wait listed patients who declined enrollment due to personal choice

SECONDARY OUTCOMES:
Sustained Virologic Response (SVR) Follow Up 1 | 24 weeks
  Among the patients who develop HCV viremia SVR rates with DAA will be measured
Sustained Virologic Response (SVR) Follow Up 2 | 48 weeks
  Among the patients who develop HCV viremia SVR rates with DAA will be measured
Liver Disease | 1 year
  Among patients who develop HCV viremia liver disease progression will be measured using non-invasive panels like fibroscan

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Gupta, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Derived] Gupta G, Yakubu I, Bhati CS, Zhang Y, Kang L, Patterson JA, Andrews-Joseph A, Alam A, Ferreira-Gonzalez A, Kumar D, Moinuddin IK, Kamal L, King AL, Levy M, Sharma A, Cotterell A, Reichman TW, Khan A, Kimball P, Stiltner R, Baldecchi M, Brigle N, Gehr T, Sterling RK. Ultra-short duration direct acting antiviral prophylaxis to prevent virus transmission from hepatitis C viremic donors to hepatitis C negative kidney transplant recipients. Am J Transplant. 2020 Mar;20(3):739-751. doi: 10.1111/ajt.15664. Epub 2019 Nov 15. PMID 31652392